CLINICAL TRIAL: NCT00098774
Title: Intensive Chemotherapy And Immunotherapy In Patients With Newly Diagnosed Primary CNS Lymphoma
Brief Title: Rituximab and Combination Chemotherapy in Treating Patients With Newly Diagnosed Primary CNS Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-50202; U10CA031946 (NIH); CALGB-50202; CDR0000398106 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma
Keywords: primary central nervous system non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Rituximab; Cytarabine; Etoposide; Leucovorin; Methotrexate; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intensive Combination Chemo & Immunotherapy (Experimental): Induction Cycles 1-3: Methotrexate 8gm/m^2 days 1 & 15; Leucovorin 100 mg/m^2 days 2 & 16; Rituximab 375 mg/m^2 days 3, 10, 17 & 24 of cycle 1, days 3 & 10 of cycle 2; Temozolomide 150 mg/m^2/day PO days 7-11
  Induction Cycle 4: Temozolomide 150 mg/m^2/day PO days 7-11; Methotrexate 8gm/m^2 day 15; Leucovorin 100 mg/m^2 day 16
  Consolidation Cycle 5: Methotrexate 8gm/m^2 days 1; Leucovorin 100 mg/m^2 days 2; Temozolomide 150 mg/m^2/day PO days 7-11
  Consolidation Cycle 6: Cytarabine 2 g/m^2 (x 8 doses) days 1-4; Etoposide 5 mg/kg (x 8 doses) days 1-4; G-CSF 5 mcg/kg/day or GM-CSF 250 mcg/m^2/day starting day 14 until ANC recovers (>= 500 for 2 consecutive days or >= 1500 for one day)
  Interventions: Biological: filgrastim; Biological: rituximab; Drug: cytarabine; Drug: etoposide; Drug: leucovorin calcium; Drug: methotrexate; Drug: temozolomide

INTERVENTIONS:
Biological: filgrastim — 5 mcg/kg subQ injection daily Day 14 until ANC > or = 500 uL for 2 days or 1500 uL for 1 day (Cycle 6)
  Other Names: G-CSF
Biological: rituximab — 375 mg/sq m IV infusion (max rate of 400 mg/hr) on Days 3, 10, 17, & 24 of Cycle 1 nad Days 3 & 10 of Cycle 2
Drug: cytarabine — 2 g/sq m IV infusion over 2 hours q 12 hrs x 8 doses Days 1-4 of Cycle 6
Drug: etoposide — 5 mg/kg IV infusion over 12 hrs q 12 hrs x 8 doses Days 1-4 of Cycle 6
Drug: leucovorin calcium — 100 mg/sq m IV infusion q 6 hrs starting 24 hrs after ea MTX dose until serum MTX < or = 0.05uM Cycles 1-5.
Drug: methotrexate — 8 g/sq m IV infusion over 4 hrs Days 1 & 15 Cycles 1, 2, & 3; Day 15 Cycle 4 and Day 1 Cycle 5.
Drug: temozolomide — 150 mg/sq m PO Days 7-11 Cycles 1-5.

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving rituximab with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase II trial is studying how well rituximab given with combination chemotherapy works in treating patients with newly diagnosed primary CNS lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete response rate after remission induction therapy with the combination of high-dose methotrexate (HDMTX), temozolomide, and rituximab at 4 months.

Secondary

* Determine the safety and feasibility of consolidation therapy comprising cytarabine and etoposide administered after induction therapy in these patients.
* Determine the percentage of patients who achieve durable (complete and partial) remission when treated with this regimen.
* Determine relapse-free survival after complete response in patients treated with this regimen.
* Correlate molecular markers with outcome in patients treated with this regimen.
* Determine the effects of this regimen on neurological function in these patients.

OUTLINE: This is a multicenter study.

* Induction Chemotherapy: All induction therapy courses repeat every 28 days.

  * Courses 1-3: Patients receive high-dose methotrexate IV over 4 hours on days 1 and 15, leucovorin calcium IV or orally every 6 hours beginning on days 2 and 16 and continuing until blood levels of methotrexate are in a safe range, and oral temozolomide on days 7-11. Patients also receive rituximab* IV on days 3, 10, 17, and 24 of course 1 and days 3 and 10 of course 2 (total of 6 doses).

NOTE: *Patients diagnosed with T-cell primary CNS lymphoma do not receive rituximab.

* Course 4: Patients receive oral temozolomide on days 7-11, high-dose methotrexate IV over 4 hours on day 15, and leucovorin calcium IV or orally every 6 hours beginning on day 16 and continuing until blood levels of methotrexate are in a safe range. Patients achieving a complete response or a complete response unconfirmed proceed to consolidation therapy.

  * Consolidation therapy I (course 5): Beginning 4 weeks after the start of course 4, patients receive high-dose methotrexate IV over 4 hours on day 1, leucovorin calcium IV or orally every 6 hours beginning on day 2 and continuing until blood levels of methotrexate are in a safe range, and oral temozolomide on days 7-11.
  * Consolidation therapy II (course 6): Beginning 3-5 weeks after the start of course 5, patients receive cytarabine IV over 2 hours twice daily and etoposide IV over 12 hours twice daily on days 1-4 and filgrastim (G-CSF) or sargramostim (GM-CSF) subcutaneously beginning on day 14 and continuing until blood counts recover.

Treatment continues in the absence of disease progression.

After completion of study treatment, patients are followed periodically for 3 years.

PROJECTED ACCRUAL: A total of 27-45 patients will be accrued for this study within 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed primary CNS lymphoma confirmed by 1 of the following methods:

  * Brain biopsy or resection
  * Cerebrospinal fluid (CSF) cytology

    * Positive CSF cytology with or without measurable intracranial disease
* No evidence of systemic non-Hodgkin's lymphoma

  * CT scan or MRI of the chest, abdomen, and pelvis AND bilateral bone marrow biopsy or unilateral biopsy with a 2cm core biopsy specimen that is negative for extracerebral source of lymphoma
* Measurable contrast-enhancing disease by MRI of the brain and spine (plus gadolinium) unless CSF cytology positive
* No evidence of pleural effusions or ascites

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3

Hepatic

* ALT and AST ≤ 2 times upper limit of normal
* Bilirubin ≤ 2 mg/dL

Renal

* Creatinine clearance ≥ 50 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 6 months after study participation
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Concurrent steroids for the management of symptoms related to lymphoma allowed

Radiotherapy

* No concurrent palliative radiotherapy

Surgery

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-10; Primary Completion 2010-01 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Rubenstein, MD, PhD, Study Chair — University of California, San Francisco
Locations (30):
- United States (30):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Union Hospital Cancer Program at Union Hospital, Elkton MD, Maryland
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Stony Brook University Cancer Center, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia

REFERENCES:
- [Result] Rubenstein JL, Hsi ED, Johnson JL, Jung SH, Nakashima MO, Grant B, Cheson BD, Kaplan LD. Intensive chemotherapy and immunotherapy in patients with newly diagnosed primary CNS lymphoma: CALGB 50202 (Alliance 50202). J Clin Oncol. 2013 Sep 1;31(25):3061-8. doi: 10.1200/JCO.2012.46.9957. Epub 2013 Apr 8. PMID 23569323

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2004 and November 2009, 47 participants were recruited at 12 CALGB sites.
Pre-assignment Details: Three participants were excluded from analysis because of failure to meet eligibility criteria or to receive protocol therapy.
Period: Overall Study
Arm/Group | Intensive Combination Chemo & Immunotherapy
Started | 44
Completed | 26
Not Completed | 18
Not completed — Adverse Event | 2
Not completed — Disease Progression | 9
Not completed — Withdrawal by Subject | 1
Not completed — Failed (to respond) during induction | 4
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intensive Combination Chemo & Immunotherapy
Number analyzed (Participants) | 44
Age, Continuous [Median (Full Range); unit: years] | 61 [12 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate After Remission Induction
Description: Response is assessed by investigator according to Revised Response Criteria for Malignant Lymphoma. Complete response requires disappearance of all evidence of disease.
Time Frame: 4 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intensive Combination Chemo & Immunotherapy
Number analyzed (Participants) | 44
percentage of participants | 66 [50 to 80]

2. Secondary Outcome: 4 Year Progression Free Rate
Description: Percentage of patients who were progression free at 4 years. The 4-year progression free rate was estimated using the Kaplan Meier method.
  Relapse was assessed by investigator according to Revised Response Criteria for Malignant Lymphoma. Progression required a 25% increase of previous area of gadolinium enhancement, appearance of new areas of T1 gadolinium enhancement or new appearance of malignant cells in the spinal fluid or new tumor appearance in other sites of the body
Time Frame: 4 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intensive Combination Chemo & Immunotherapy
Number analyzed (Participants) | 44
percentage of participants | 48 [33 to 63]

3. Secondary Outcome: Change From Baseline in Mini-Mental Status Evaluation at 4 Months
Description: Neurologic functioning will be assessed using the Mini-Mental Status Evaluation (MMSE), a standardized, bedside tool for evaluation of higher mental function. This assessment is based on a 30-point scale (0-30) with higher scores associated with better performance.
Time Frame: Baseline & month 4
Population: Only 14 participants had both baseline and 4 month MMSE evaluations reported.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Intensive Combination Chemo & Immunotherapy
Number analyzed (Participants) | 14
units on a scale
  Baseline Score | 27 [7 to 30]
  4 month Score | 28 [22 to 30]
  Change from Baseline | 1 [-1 to 18]

4. Secondary Outcome: 4 Year Overall Survival Rate
Description: Percentage of patients who were alive at 4 years. The 4-year survival rate was estimated using the Kaplan Meier method.
Time Frame: 4 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intensive Combination Chemo & Immunotherapy
Number analyzed (Participants) | 44
percentage of participants | 65 [49 to 77]

ADVERSE EVENTS:
Arm/Group | Intensive Combination Chemo & Immunotherapy
Serious Adverse Events (participants affected / at risk) | 15/44
Other Adverse Events (participants affected / at risk) | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive Combination Chemo & Immunotherapy (N=44)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 11 (13)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 3 (3)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 7 (7)
Rectal mucositis (Gastrointestinal disorders) | 2 (2)
Small intestinal mucositis (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5)
Chills (General disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 7 (7)
Fever (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Anorectal infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Lymph gland infection (Infections and infestations) | 1 (1)
Opportunistic infection (Infections and infestations) | 1 (1)
Peritoneal infection (Infections and infestations) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 8 (10)
Alkaline phosphatase increased (Investigations) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 7 (8)
Blood bilirubin increased (Investigations) | 6 (6)
Creatinine increased (Investigations) | 4 (4)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
Laboratory test abnormal (Investigations) | 3 (3)
Leukocyte count decreased (Investigations) | 6 (6)
Lymphocyte count decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 9 (10)
Platelet count decreased (Investigations) | 10 (10)
Serum cholesterol increased (Investigations) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Blood glucose increased (Metabolism and nutrition disorders) | 10 (10)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 6 (6)
Serum calcium decreased (Metabolism and nutrition disorders) | 6 (6)
Serum magnesium decreased (Metabolism and nutrition disorders) | 4 (4)
Serum magnesium increased (Metabolism and nutrition disorders) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 7 (7)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 3 (3)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (Nervous system disorders) | 3 (4)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Intracranial hemorrhage (Nervous system disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 3 (5)
Mini mental status examination abnormal (Nervous system disorders) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 3 (3)
Nystagmus (Nervous system disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 4 (5)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (3)
Hypertension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 4 (4)
Vascular disorder (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive Combination Chemo & Immunotherapy (N=44)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7)
Hemoglobin decreased (Blood and lymphatic system disorders) | 30 (90)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 2 (4)
Edema (Cardiac disorders) | 1 (3)
Palpitations (Cardiac disorders) | 2 (3)
Sinus bradycardia (Cardiac disorders) | 3 (4)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 2 (3)
Cushingoid (Endocrine disorders) | 1 (1)
Diplopia (Eye disorders) | 2 (5)
Dry eye syndrome (Eye disorders) | 2 (2)
Eye disorder (Eye disorders) | 3 (4)
Eye pain (Eye disorders) | 1 (1)
Flashing vision (Eye disorders) | 3 (3)
Keratitis (Eye disorders) | 1 (3)
Photophobia (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 7 (16)
Watering eyes (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 19 (37)
Diarrhea (Gastrointestinal disorders) | 23 (45)
Dry mouth (Gastrointestinal disorders) | 1 (6)
Dyspepsia (Gastrointestinal disorders) | 6 (7)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 16 (22)
Nausea (Gastrointestinal disorders) | 36 (92)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT studies, if specified in (Gastrointestinal disorders) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 25 (44)
Chest pain (General disorders) | 3 (3)
Chills (General disorders) | 6 (7)
Edema limbs (General disorders) | 16 (36)
Fatigue (General disorders) | 32 (83)
Fever (General disorders) | 8 (9)
General symptom (General disorders) | 2 (2)
Localized edema (General disorders) | 1 (3)
Pain (General disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 2 (3)
Bladder infection (Infections and infestations) | 2 (2)
Catheter related infection (Infections and infestations) | 3 (4)
Eye infection (Infections and infestations) | 1 (1)
Gingival infection (Infections and infestations) | 2 (3)
Infection (Infections and infestations) | 4 (4)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 1 (1)
Infectious colitis (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Opportunistic infection (Infections and infestations) | 1 (1)
Phlebitis infective (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Upper aerodigestive tract infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (6)
Vaginal infection (Infections and infestations) | 1 (3)
Wound infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 32 (85)
Alkaline phosphatase increased (Investigations) | 8 (11)
Aspartate aminotransferase increased (Investigations) | 33 (81)
Blood bilirubin increased (Investigations) | 20 (32)
Creatinine increased (Investigations) | 17 (32)
Fibrinogen decreased (Investigations) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (3)
Laboratory test abnormal (Investigations) | 5 (7)
Leukocyte count decreased (Investigations) | 14 (39)
Lymphocyte count decreased (Investigations) | 3 (7)
Neutrophil count decreased (Investigations) | 31 (59)
Platelet count decreased (Investigations) | 30 (52)
Serum cholesterol increased (Investigations) | 2 (3)
Weight gain (Investigations) | 2 (3)
Weight loss (Investigations) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 19 (43)
Blood glucose increased (Metabolism and nutrition disorders) | 19 (53)
Blood uric acid increased (Metabolism and nutrition disorders) | 4 (6)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Serum albumin decreased (Metabolism and nutrition disorders) | 20 (41)
Serum calcium decreased (Metabolism and nutrition disorders) | 14 (32)
Serum glucose decreased (Metabolism and nutrition disorders) | 3 (5)
Serum magnesium decreased (Metabolism and nutrition disorders) | 7 (13)
Serum magnesium increased (Metabolism and nutrition disorders) | 2 (4)
Serum phosphate decreased (Metabolism and nutrition disorders) | 4 (9)
Serum potassium decreased (Metabolism and nutrition disorders) | 26 (68)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 15 (32)
Serum sodium increased (Metabolism and nutrition disorders) | 4 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 8 (13)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4)
Ataxia (Nervous system disorders) | 15 (19)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 10 (11)
Dysgeusia (Nervous system disorders) | 5 (10)
Encephalopathy (Nervous system disorders) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (6)
Headache (Nervous system disorders) | 21 (47)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 6 (12)
Mini mental status examination abnormal (Nervous system disorders) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 3 (3)
Nystagmus (Nervous system disorders) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 7 (17)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (21)
Seizure (Nervous system disorders) | 4 (5)
Speech disorder (Nervous system disorders) | 3 (4)
Syncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 3 (3)
Trigeminal nerve disorder (Nervous system disorders) | 1 (6)
Anxiety (Psychiatric disorders) | 11 (20)
Confusion (Psychiatric disorders) | 13 (19)
Depression (Psychiatric disorders) | 8 (16)
Insomnia (Psychiatric disorders) | 9 (25)
Psychosis (Psychiatric disorders) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (2)
Urogenital disorder (Renal and urinary disorders) | 3 (5)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (19)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (4)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7)
Rash desquamating (Skin and subcutaneous tissue disorders) | 21 (27)
Skin disorder (Skin and subcutaneous tissue disorders) | 3 (4)
Hemorrhage (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 8 (13)
Hypotension (Vascular disorders) | 4 (4)
Phlebitis (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less